CLINICAL TRIAL: NCT05368246
Title: Safety and Performance of UCon for the Treatment of the Symptoms of Overactive Bladder (OAB) / Bowel Dysfunction (BD) - An Early Feasibility Study
Brief Title: Safety and Performance of UCon for the Treatment of the Symptoms of Overactive Bladder (OAB) / Bowel Dysfunction (BD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnoCon Medical (Industry)
Collaborators: Aarhus University Hospital (Other); Herlev Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK_FEAS_01
Record Dates: First submitted 2022-04-25; First posted 2022-05-10 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Urinary Incontinence; Fecal Incontinence; Urge Incontinence; Nocturia; Urinary Frequency More Than Once at Night; Bowel Disorders Functional; Urinary Incontinence, Urge; Incontinence, Nighttime Urinary
Keywords: Urinary Incontinence; Fecal Incontinence; Urge incontinence; Neurostimulation; Dorsal Genital Nerve; Nocturia
MeSH Terms: conditions — Urinary Incontinence; Fecal Incontinence; Urinary Incontinence, Urge; Nocturia; Nocturnal Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Electrical stimulation to the dorsal genital nerve.
  Interventions: Device: UCon

INTERVENTIONS:
Device: UCon — The subjects self-administer electrical stimulation to the dorsal genital nerve (DGN) for 4 weeks using UCon

SUMMARY:
This clinical investigation is a single-arm, prospective, multicentre, early feasibility study, which is used to evaluate the device design of UCon with respect to initial clinical safety and device performance in a small number of subjects. UCon is a medical device for treatment of the symptoms of overactive bladder (OAB) and bowel disorders (BD). It electrically stimulates the dorsal genital nerve (DGN) through the skin to obtain modulated behaviour of the bladder/bowel musculature e.g., suppress undesired bladder/bowel activity to relieve the symptoms of the patient.

DETAILED DESCRIPTION:
The study is conducted at multiple hospitals in Denmark (Aarhus University Hospital, Odense University Hospital and Herlev Hospital). It is estimated that 20 subjects with OAB and 20 subjects with BD will need to be enrolled at the investigational sites to account for screening attrition and dropouts. Screening and baseline measurements includes a 7-days bladder diary (OAB) / 14-days bowel diary (BD) and quality-of-life measures. Following the screening and baseline measurements, the subjects will be introduced and trained on how to set up and use UCon. For 1 month the subjects will use UCon at home and complete a daily bladder/bowel diary and a stimulation diary. After completion of the interventional period, subjects will fill out the quality-of-life measures once again.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject is diagnosed with OAB or BD.
3. Subject is able to communicate, provide feedback, understand and follow instructions during the course of the study.
4. Subject has signed an informed consent.

Exclusion Criteria:

1. Subject is medically unstable.
2. Subject has an active infection in the genital area.
3. Subject has an implanted pacemaker, implantable drug pump or other active medical device (any medical device that uses electrical energy or other source of power to make it function).
4. Subject is pregnant, nursing or planning a pregnancy (to be confirmed with a negative pregnancy test within 14 days prior to enrolment). Women of childbearing potential must maintain effective contraception* during the study period judged by the investigator.
5. Subject is enrolled or planning to enrol in another investigational study or was enrolled in an investigational drug or medical device trial within four weeks to enrolment.
6. Subject has neuropathy to a degree that is presumed to diminish the effect of the electrical stimulation.
7. Subject has a history of cancer in the pelvic region, are currently receiving cancer treatment, or has radiation-induced damage to the pelvic region.
8. Subject has addictive behaviour defined as abuse of cannabis, opioids, or other intoxicating drugs.
9. Subject does not speak and understand Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Characterization of adverse events related to the risks and anticipated adverse device effects associated with the use of UCon. | After 4 and 12 weeks of stimulation (end of study).
  Characterization of adverse events related to the risks and anticipated adverse device effects associated with the use of UCon during the study period.
Ratio of subjects with at least 50% improvement of their OAB/BD symptoms from baseline associated with the use of UCon. | Change from baseline OAB/BD symptoms at 4 and 12 weeks.
  Urinary urgency is measured by number of urgency episodes/day. Urinary frequency is measured by number of voidings/day. Urgency urinary incontinence is measured by number of leaks preceded by urgency/day.
  Nocturia is measured by number of voidings/night. Faecal urgency is measured by number of urgency episodes/day. Frequent bowel movements are measured by number of voidings/day. Faecal incontinence (urge/passive) is measured by number of leaks/day.

SECONDARY OUTCOMES:
Frequency and severity of all adverse events related to the risks and anticipated adverse device effects associated with the use of UCon. | After 4 and 12 weeks of stimulation (end of study).
  Number of subjects experiencing adverse events related to the risks and anticipated adverse device effects associated with the use of UCon during the study period.
  Number and severity of adverse events related to the risks and anticipated adverse device effects associated with the use of UCon during the study period.
Ratio of subjects with improvement in their OAB/BD specific quality-of-life measures from baseline. | Change from baseline QoL at 4 and 12 weeks.
  For OAB the following is used to assess QoL: "International Consultation on Incontinence Questionnaire Overactive Bladder Module". It contains 4 questions and a higher total score means a worse outcome.
  For BD a combination of the following is used to assess QoL: "St. Marks incontinence score" and "Rockwood Fecal Incontinence Quality of Life Scale". St. Marks incontinence score contains 7 questions, and a higher total score means a worse outcome. The Rockwood Fecal Incontinence Quality of Life Scale contains 29 questions and a higher total score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Christensen, Principal Investigator — Palle Juul Jensens Boulevard 99 DK-8200 Aarhus N
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus, Aarhus N
  - Herlev Hospital, Herlev, Region Sjælland
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grau LS, Christensen P, Qvist N, Klarskov N, Rijkhoff N, Duelund-Jakobsen J. Dorsal Genital Nerve Stimulation in Patients With Fecal Incontinence and Fecal Urgency: A Feasibility Study With the Novel UCon Neurostimulator. Neurogastroenterol Motil. 2025 Dec 20:e70225. doi: 10.1111/nmo.70225. Online ahead of print. PMID 41420462